CLINICAL TRIAL: NCT01938365
Title: A Prospective Cohort Study of Clinical Characteristics and Genetic Susceptibility of Type 1 Diabetes in Chinese Adolescents and Youth
Brief Title: Genetics of Type 1 Diabetes in Chinese Adolescents and Youth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Professor, Shanghai Jiao Tong University School of Medicine
Other Study IDs: CCEMD020
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood,fasting serum and stool
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetes
- Normal glucose regulation

SUMMARY:
primary outcome: To explore the genetic susceptibility of diabetes in Chinese adolescent and youth.

secondary outcomes:

1. To classify diabetes by gene detection in Chinese adolescent and youth.
2. To make the relationship between genotype and clinic phenotype in type 1 diabetes.
3. To evaluate the effect of environmental factors (intestinal ecosystem)in the pathogenesis of diabetes.

DETAILED DESCRIPTION:
Phase 1: Baseline investigation Aims: To explore genetic susceptibility of diabetes in Chinese adolescent and youth.

Subjects and Methods: 500 patients under diabetic conditions and sex,age-matched NGR Healthy control(2:1) will be enrolled ,all aged from 14-30 years old. A comprehensive examination including questionnaire, anthropometric measurements, biochemical analysis will be performed in each study participant. Diabetes should be diagnosed according to the WHO 1999 criteria,type 1 or type 2 diabetes diagnosed by clinical features recommended by International Society of Pediatric and Adolescent Diabetes ( ISPAD ).

Phase 2: Cohort follow-up Aims : To explore the association of genetic backgrounds and clinical characteristics in different types of diabetes in Chinese adolescent and youth.

Subjects and Methods: To recruit and follow up 200 newly diagnosed and genotyped patients for 3 years. Questionnaire, anthropometric measurements, biochemical analysis performed respectively at baseline,3,6,12,24,36 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 14- 30 years old
2. Gender: males and females
3. Race: han
4. Diabetes diagnosed by WHO cafeteria (WHO1999)
5. Living in east China area to minimize population stratification

Exclusion Criteria:

1. Secondary diabetes caused by other diseases or drugs
2. Moderate to severe liver, kidney dysfunction, i.e. ALT/AST > 2.5 times the upper limit of normal range or Ccr < 25ml/min;
3. Any other condition or major systemic diseases that the investigator feels would interfere with trial participation or evaluation of results.

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: In phase 1:500 patients under diabetic conditions and sex,age-matched NGR(Normal glucose regulation) (2:1) will be enrolled ,all aged from 14-30.
  In phase 2:200 patients newly diagnosed diabetes (less than 6 month before enrollment )will be genotyped and followed up for 3 years
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Deterioration of pancreatic islet function | 3 years

SECONDARY OUTCOMES:
Insulin dosage, HbA1c levels and evaluation of chronic complications | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Gao A, Gu B, Zhang J, Fang C, Su J, Li H, Han R, Ye L, Wang W, Ning G, Wang J, Gu W. Missense Variants in PAX4 Are Associated with Early-Onset Diabetes in Chinese. Diabetes Ther. 2021 Jan;12(1):289-300. doi: 10.1007/s13300-020-00960-5. Epub 2020 Nov 20. PMID 33216280